CLINICAL TRIAL: NCT02188147
Title: Ambulatory Post-Syncope Arrhythmia Protection Feasibility Study Protocol
Brief Title: Ambulatory Post-Syncope Arrhythmia Protection Feasibility Study
Acronym: ASAP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Zoll Medical Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 90D0119
Record Dates: First submitted 2014-07-09; First posted 2014-07-11 (Estimated); Results first posted 2023-02-21 (Actual); Last update posted 2023-02-21 (Actual); Status verified 2023-01

CONDITIONS: Syncope
Keywords: Syncope; Sudden Cardiac Arrest; Sudden Cardiac Death; Cardiac Arrest; Emergency Service; Emergency Department; Ambulatory Electrocardiography; Holter; Holter Electrocardiography; Holter Monitoring
MeSH Terms: conditions — Syncope; Death, Sudden, Cardiac; Heart Arrest; Emergencies

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- SWD 1000 (Experimental): Short Term Wearable Defibrillator
  Interventions: Device: Short Term Wearable Defibrillator

INTERVENTIONS:
Device: Short Term Wearable Defibrillator — Short-term Wearable Defibrillator (SWD 1000)

SUMMARY:
The purpose of this study is to conduct an observational investigation of a novel care path used to manage emergency department (ED) presenting syncope patients on an outpatient basis.

DETAILED DESCRIPTION:
OBJECTIVES To conduct a prospective observational study assessing a unique outpatient care model in which syncope patients are provided with, and trained to use, a wearable defibrillator prior to discharge from the emergency department (ED). Observational data will be collected to assess the logistics of equipping patients with the device and providing training in the ED, and the ability of patients to receive follow-up care on an outpatient basis. In addition, data will be collected to confirm that the device meets expected safety. The experience gained from this stage of the study will be used to guide future studies of device's functionality enhancements and definitive device safety and efficacy.

STUDY POPULATION Participants will be patients presenting to the ED following a syncope event which has been defined as cardiac, or potentially cardiac, i.e. undiagnosed in nature.

INTERVENTION A wearable defibrillator optimized for short-term ambulatory use with adhesive electrodes will be prescribed for up to 14 days of use following emergency department discharge or until the physician responsible for the subject's care defines an alternative treatment plan.

STUDY DESIGN This is a single-arm feasibility study.

STUDY SIZE The study will enroll a minimum of 50 and a maximum of 80 subjects. A maximum of 20 centers will be used for enrollment.

ELIGIBILITY:
Inclusion Criteria:

1. Age≥18
2. Experienced a syncopal event within the past 48 hours
3. Either one of the following profiles(A or B) apply:

A. ED workup indicates that the patient may have experienced syncope that is cardiac in nature (any one or more of the following apply:

* History or diagnosis of structural heart disease
* History of cardiovascular disease
* Age ≥ 40
* Palpitations experienced pre-syncope
* Major ECG abnormalities:

  * QRS-duration greater than 140 ms
  * PR-interval greater than 200 ms
  * Non-specific repolarization abnormality
* Syncope experienced without any warning
* Syncope experienced while supine
* Syncope during exercise B. ED workup does not indicate a clear cause of the syncopal event

Exclusion Criteria:

1. Clear diagnosis of non-cardiac syncope (e.g. orthostatic hypotensive syncope, vasovagal syncope, carotid sinus syncope, situational fainting)
2. An active implantable cardioverter-defibrillator (ICD)
3. An active unipolar pacemaker
4. Significant risk or suffering a cardiovascular event such as:

   * Symptoms of New York Heart Association (NYHA) class III or IV heart failure
   * ED diagnosis of acute coronary syndrome
   * Having required resuscitation in response to the index syncopal event
   * Advanced directive prohibiting resuscitation (DNR)

6. Physical or mental conditions preventing subjects from interacting with or wearing the device as determined by the investigating physician.

7. Bandages or other clinical condition preventing SWD 1000 use 8. Injuries or other conditions beyond simple syncope that require hospitalization 9. Travel out of town during the study participation period that prevents the field service representative from visiting the subject daily 10. Unable or unwilling to provide written informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2014-08 (Actual); Primary Completion 2020-04 (Actual); Study Completion 2020-04-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Steve Szymkiewicz, MD, Study Director — Zoll Medical Corporation
Locations (6):
- United States (6):
  - Danbury, Connecticut
  - Jacksonville, Florida
  - Minneapolis, Minnesota
  - Saint Paul, Minnesota
  - Staten Island, New York
  - Cincinnati, Ohio

RESULTS

PARTICIPANT FLOW:
Groups:
- SWD 1000: Patients who presented to the emergency room after syncope, and their syncopal event was believed to have a cardiac or undiagnosed cause. In this group participants agreed to wear the Short Term Wearable Defibrillator 1000 (SWD 1000) after discharge for up to 14 days.
Period: Overall Study
Arm/Group | SWD 1000
Started | 39
Completed | 39
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- SWD 1000: Subjects assigned to use a Short Term Wearable Defibrillator (SWD 1000)
Arm/Group | SWD 1000
Number analyzed (Participants) | 39
Age, Continuous [Mean (Standard Deviation); unit: years] | 44.4 (17.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15
  Male | 24
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 0
  Unknown or Not Reported | 39
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 0
  More than one race | 0
  Unknown or Not Reported | 39
Height [Mean (Standard Deviation); unit: inches] | 67.5 (3.8)
Weight [Mean (Standard Deviation); unit: pounds] | 185.2 (51.6)
Blood pressure [Mean (Standard Deviation); unit: mm Hg]
  Systolic | 127 (18)
  Diastolic | 76 (13)
Heart rate [Mean (Standard Deviation); unit: beats per minute] | 76 (15)
Respiration rate [Mean (Standard Deviation); unit: breaths per minute] | 16.4 (2.5)
Prior syncope [Count of Participants; unit: Participants] | 29
Past history of myocardial infarction [Count of Participants; unit: Participants] | 3
Past history of heart failure [Count of Participants; unit: Participants] | 3
Past history of diabetes [Count of Participants; unit: Participants] | 9
Past history of atrial fibrillation [Count of Participants; unit: Participants] | 2
Past history of renal failure [Count of Participants; unit: Participants] | 1
Active pacemaker [Count of Participants; unit: Participants] | 1
Family history of sudden death [Count of Participants; unit: Participants] | 6

OUTCOME MEASURES:

1. Primary Outcome: Device Unable to Monitor Due to ECG Noise
Description: % time the device detected noise on both leads at the same time.
Time Frame: enrollment to 30 days
Population: Subjects who used the SWD1000 for at least 24 hours
Measure: Mean (90% Confidence Interval); unit: percentage of time worn
Arm/Group | SWD 1000
Number analyzed (Participants) | 30
percentage of time worn | 1.5 [0.59 to 2.39]

2. Primary Outcome: Device Monitoring Using Only One ECG Lead
Description: % time that the device is monitoring using only one lead due to noise detected on the other lead
Time Frame: enrollment to 30 days
Population: SWD 1000 participants who used the device at least 24 hours.
Measure: Mean (90% Confidence Interval); unit: percentage of time worn
Arm/Group | SWD 1000
Number analyzed (Participants) | 30
percentage of time worn | 2.5 [2.44 to 4.18]

3. Primary Outcome: Followup Care Visits
Description: Followup care for syncope - outpatient medical care visits
Time Frame: enrollment to 30 days
Measure: Count of Participants; unit: Participants
Arm/Group | SWD 1000
Number analyzed (Participants) | 39
Participants | 17

4. Primary Outcome: ER or Hospitalization
Description: Followup care for syncope - returned to ER or admitted to hospital
Time Frame: enrollment to 30 days
Measure: Count of Participants; unit: Participants
Arm/Group | SWD 1000
Number analyzed (Participants) | 39
Participants | 4

5. Secondary Outcome: Duration of Use
Description: Average time the SWD 1000 was used by participants
Time Frame: enrollment to 30 days
Measure: Mean (Standard Deviation); unit: days
Arm/Group | SWD 1000
Number analyzed (Participants) | 39
days | 6.1 (5.2)

6. Post Hoc Outcome: Noise Alarms
Description: SWD 1000 alarms given to alert user of detected noise on one or more ECG leads
Time Frame: enrollment to 30 days
Measure: Mean (Standard Deviation); unit: count of alarms per subject
Arm/Group | SWD 1000
Number analyzed (Participants) | 39
count of alarms per subject | 15 (17)

7. Post Hoc Outcome: Arrhythmia Alarms
Description: Device alarms given because an arrhythmia was detected (may or may not be real arrhythmia)
Time Frame: enrollment to 30 days
Measure: Mean (Standard Deviation); unit: number of alarms per subjects
Arm/Group | SWD 1000
Number analyzed (Participants) | 39
number of alarms per subjects | 9.9 (31.1)

ADVERSE EVENTS:
Time Frame: 30 days
Arm/Group | SWD 1000
All-Cause Mortality (participants affected / at risk) | 0/39
Serious Adverse Events (participants affected / at risk) | 0/39
Other Adverse Events (participants affected / at risk) | 13/39
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | SWD 1000 (N=39)
Skin rash or irritation (Skin and subcutaneous tissue disorders) | 10 (12) — Skin rash or irritation (no medical intervention required)
Inappropriate shock (Injury, poisoning and procedural complications) | 3 (3) — A defibrillation shock was delivered when the patient was not experiencing a treatable arrhythmia

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-01-15): https://cdn.clinicaltrials.gov/large-docs/47/NCT02188147/Prot_SAP_000.pdf